CLINICAL TRIAL: NCT01365975
Title: Follow-up Study of Late Effects of Periconceptional Folic Acid in Mothers and Offspring in the Community Intervention Program Population: The Chinese Children and Families Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911165; 11-C-N165
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Pediatric Leukemia; Other Pediatric Cancers
Keywords: Cohort Study; Folic Acid Peri-Conception; Pediatric Leukemia; Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Community Intervention Program Population: The Chinese Childre: Community sample of mothers, fathers and offspring from 2 provinces in China who participated in a community public health study in 1994-1996.

SUMMARY:
Periconceptional folic acid supplements of 400 (Micro) daily prevent neural tube defects (NTD) in offspring. Some data suggest that periconceptional folic acid supplements, folate levels during pregnancy, and/or certain variants in the gene that encodes methylenetetrahydrofolate reductase (MTHFR), a key enzyme that catalyzes synthesis of 5-methyltetrahydrofolate [the primary methyl donor in most metabolic pathways involving methylation including DNA methylation] from 5,10 methylenetetrahydrofolate may be associated with reduced risks of certain adverse events during the prenatal period, birth weight and certain serious diseases in offspring, while other studies have raised concerns about increased risks of specific serious disorders. Only one study has examined late health effects in mothers that might be associated with use of periconceptional folic acid supplements.

We propose to study potential health benefits and adverse effects of periconceptional folic acid supplements in a 15-year follow-up of offspring and mothers. In the offspring, we will evaluate whether periconceptional folic acid supplements reduced risk of external congenital birth defects and childhood acute lymphoblastic leukemia, and whether risks are reduced or increased for other pediatric disorders linked with periconceptional folic acid supplements including asthma, pervasive developmental disorders and autism, diabetes, obesity and blood pressure. In the mothers, we will assess cardiovascular diseases and associated risk factors, breast and colorectal cancers and precursor conditions, and other cancers. We will also conduct exploratory assessment of other serious diseases in mothers.

To increase the limited data on the morbidity and survival of children born with a major birth defect, particularly in low- or middle-income countries, we plan to assess morbidity and mortality outcomes in children identified with neural tube defects as part of our follow-up.

The women and children who participated in the joint China-U.S. Community Intervention Program (CIP) trial (N=243,779 women treated or not treated with folic acid in the periconceptional period and their offspring) represent unique cohorts whose periconceptional exposure to folic acid is well documented. We propose to follow a sample of 22,000 CIP mothers and their offspring (currently 14 to 17 years of age), to ascertain vital status, medical history, and lifestyle habits. The study will clarify whether there are differences with respect to growth, physical development during the puberty period, selected serious morbidity and mortality in offspring and risks of serious health outcomes and mortality in mothers associated with periconceptional folic acid supplements. Data from this study will inform us about cohort participation rate, cost, and effective approaches for future follow-up of the full cohort.

The current protocol focuses on a pilot study (Pilot Study # 1) in which we will carry out two specific aims in 500 families. We will test and evaluate the most effective approaches to trace the mothers who enrolled in the CIP in 1993-1995 in CIP counties, fathers, and children. If the child is not living with the biological mother, we will trace the caretaker or next of kin with whom the child is living. We will also conduct in-person interviews, obtain anthropometric and blood pressure measurements and determine cohort participation rate in a sample of 500 CIP families from two of the 21 CIP project counties to obtain health information, medical history, and vital status. We will attempt to enroll in the pilot study 500 mothers/caretakers and 500 offspring, and 500 fathers (Total N=1500). Excluded from the Pilot Study #1 at this time are the families in which the mother or the child is deceased. We will seek permission from the IRB to enroll these families at a later date.

DETAILED DESCRIPTION:
Periconceptional folic acid supplements of 400 (Micro) daily prevent neural tube defects (NTD) in offspring. Some data suggest that periconceptional folic acid supplements, folate levels during pregnancy, and/or certain variants in the gene that encodes methylenetetrahydrofolate reductase (MTHFR), a key enzyme that catalyzes synthesis of 5-methyltetrahydrofolate [the primary methyl donor in most metabolic pathways involving methylation including DNA methylation] from 5,10 methylenetetrahydrofolate may be associated with reduced risks of certain adverse events during the prenatal period, birth weight and certain serious diseases in offspring, while other studies have raised concerns about increased risks of specific serious disorders. Only one study has examined late health effects in mothers that might be associated with use of periconceptional folic acid supplements.

We propose to study potential health benefits and adverse effects of periconceptional folic acid supplements in a 15-year follow-up of offspring and mothers. In the offspring, we will evaluate whether periconceptional folic acid supplements reduced risk of external congenital birth defects and childhood acute lymphoblastic leukemia, and whether risks are reduced or increased for other pediatric disorders linked with periconceptional folic acid supplements including asthma, pervasive developmental disorders and autism, diabetes, obesity and blood pressure. In the mothers, we will assess cardiovascular diseases and associated risk factors, breast and colorectal cancers and precursor conditions, and other cancers. We will also conduct exploratory assessment of other serious diseases in mothers.

To increase the limited data on the morbidity and survival of children born with a major birth defect, particularly in low- or middle-income countries, we plan to assess morbidity and mortality outcomes in children identified with neural tube defects as part of our follow-up.

The women and children who participated in the joint China-U.S. Community Intervention Program (CIP) trial (N=243,779 women treated or not treated with folic acid in the periconceptional period and their offspring) represent unique cohorts whose periconceptional exposure to folic acid is well documented. We propose to follow a sample of 22,000 CIP mothers and their offspring (currently 14 to 17 years of age), to ascertain vital status, medical history, and lifestyle habits. The study will clarify whether there are differences with respect to growth, physical development during the puberty period, selected serious morbidity and mortality in offspring and risks of serious health outcomes and mortality in mothers associated with periconceptional folic acid supplements. Data from this study will inform us about cohort participation rate, cost, and effective approaches for future follow-up of the full cohort.

The current protocol focuses on a pilot study (Pilot Study # 1) in which we will carry out two specific aims in 500 families. We will test and evaluate the most effective approaches to trace the mothers who enrolled in the CIP in 1993-1995 in CIP counties, fathers, and children. If the child is not living with the biological mother, we will trace the caretaker or next of kin with whom the child is living. We will also conduct in-person interviews, obtain anthropometric and blood pressure measurements and determine cohort participation rate in a sample of 500 CIP families from two of the 21 CIP project counties to obtain health information, medical history, and vital status. We will attempt to enroll in the pilot study 500 mothers/caretakers and 500 offspring, and 500 fathers (Total N=1500). Excluded from the Pilot Study #1 at this time are the families in which the mother or the child is deceased. We will seek permission from the IRB to enroll these families at a later date.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 500 Chinese mothers, fathers and their child aged 14-16 years
* Participated in the Community Intervention Program from 1993 to 1996
* Living in Laoting and Tai(SqrRoot)(Beta)ang Counties
* Provide consent
* The mother and child to provide answers to at least some of the questions about himself/herself and for the mother to answer some questions about the child

EXCLUSION CRITERIA:

* Not having been a singleton birth
* Missing data on pill usage
* Missing data on gender

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample of mothers, fathers and offspring from 2 provinces in China who participated in a community public health study in 1994-1996.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 1382 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of long term health effects | 1994-2012
  observational study inquiring about various measures of health including cancer, hypertension, and diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Potischman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bailey LB, Gregory JF 3rd. Folate metabolism and requirements. J Nutr. 1999 Apr;129(4):779-82. doi: 10.1093/jn/129.4.779. PMID 10203550
- [Background] Laurence KM, James N, Miller MH, Tennant GB, Campbell H. Double-blind randomised controlled trial of folate treatment before conception to prevent recurrence of neural-tube defects. Br Med J (Clin Res Ed). 1981 May 9;282(6275):1509-11. doi: 10.1136/bmj.282.6275.1509. PMID 6786536
- [Background] Smithells RW, Nevin NC, Seller MJ, Sheppard S, Harris R, Read AP, Fielding DW, Walker S, Schorah CJ, Wild J. Further experience of vitamin supplementation for prevention of neural tube defect recurrences. Lancet. 1983 May 7;1(8332):1027-31. doi: 10.1016/s0140-6736(83)92654-5. PMID 6133069